CLINICAL TRIAL: NCT00672984
Title: A Phase I, Randomized, Gender Stratified, Double-Blind, Placebo- and Positive-Controlled, Three Period Crossover Trial to Assess the Effect of Guanfacine Hydrochloride on QT/QTc Interval in Healthy Men and Women
Brief Title: Guanfacine Immediate-release Electrocardiogram Results (QTc) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPD503-112
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: QT/QTc
MeSH Terms: interventions — Guanfacine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Immediate-release Guanfacine HCl (Experimental)
  Interventions: Drug: immediate release guanfacine hydrochloride
- Moxifloxacin HCl (Active Comparator)
  Interventions: Drug: moxifloxacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: immediate release guanfacine hydrochloride — Subjects will receive 2x2mg immediate-release guanfacine on day 1. Subjects will receive 4x2mg immediate-release guanfacine on day 6.
  Other Names: Tenex
  Arms: Immediate-release Guanfacine HCl
Drug: moxifloxacin — Subjects will receive 400mg of moxifloxacin on day 1. Subjects will receive 400mg of moxifloxacin on day 6.
  Other Names: Avelox
  Arms: Moxifloxacin HCl
Drug: Placebo — Subjects will receive placebo on Day 1. Subjects will receive placebo on Day 6.
  Arms: Placebo

SUMMARY:
To assess the effect of immediate-release guanfacine hydrochloride, administered at therapeutic and supratherapeutic doses, on QT/QTc in healthy normal males and females

ELIGIBILITY:
Inclusion Criteria:

* Healthy Normal Subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2008-04-18 (Actual); Primary Completion 2008-08-07 (Actual); Study Completion 2008-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Charles River Clinical Services Northwest, Inc., Tacoma, Washington, United States

REFERENCES:
- [Derived] Martin P, Satin L, Kahn RS, Robinson A, Corcoran M, Purkayastha J, Youcha S, Ermer JC. A thorough QT study of guanfacine. Int J Clin Pharmacol Ther. 2015 Apr;53(4):301-16. doi: 10.5414/CP202065. PMID 25109412
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a three period crossover trial.
Groups:
- Guanfacine First: Single 4 mg dose of immediate-release Guanfacine HCl on Day 1, 4 mg of immediate-release Guanfacine HCl bid on Days 2 and 3, 6 mg of immediate-release Guanfacine HCl bid on Days 4 and 5, and a single 8 mg dose of immediate-release Guanfacine HCl on Day 6 in first intervention period; single 400 mg dose of Moxifloxacin on Day 1, placebo bid on Days 2, 3, 4, and 5, and single 400 mg dose of Moxifloxacin on Day 6 in second intervention period (after washout period); single dose of placebo on Day 1, placebo bid on Days 2, 3, 4, and 5, and single dose of placebo on Day 6 in third intervention period (after washout period).
- Moxifloxacin First: Single 400 mg dose of Moxifloxacin on Day 1, placebo bid on Days 2, 3, 4, and 5, and single 400 mg dose of Moxifloxacin on Day 6 in first intervention period; single dose of placebo on Day 1, placebo bid on Days 2, 3, 4, and 5, and single dose of placebo on Day 6 in second intervention period (after washout period); single 4 mg dose of immediate-release Guanfacine HCl on Day 1, 4 mg of immediate-release Guanfacine HCl bid on Days 2 and 3, 6 mg of immediate-release Guanfacine HCl bid on Days 4 and 5, and a single 8 mg dose of immediate-release Guanfacine HCl on Day 6 in third intervention period (after washout period).
- Placebo First: Single dose of placebo on Day 1, placebo bid on Days 2, 3, 4, and 5, and single dose of placebo on Day 6 in first intervention period; single 4 mg dose of immediate-release Guanfacine HCl on Day 1, 4 mg of immediate-release Guanfacine HCl bid on Days 2 and 3, 6 mg of immediate-release Guanfacine HCl bid on Days 4 and 5, and a single 8 mg dose of immediate-release Guanfacine HCl on Day 6 in second intervention period (after washout period); single 400 mg dose of Moxifloxacin on Day 1, placebo bid on Days 2, 3, 4, and 5, and single 400 mg dose of Moxifloxacin on Day 6 in third intervention period (after washout period).
Period: First Intervention
Arm/Group | Guanfacine First | Moxifloxacin First | Placebo First
Started | 31 | 25 | 27
Completed | 22 | 23 | 25
Not Completed | 9 | 2 | 2
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Sponsor decision | 3 | 0 | 0
Period: Second Intervention
Arm/Group | Guanfacine First | Moxifloxacin First | Placebo First
Started | 22 | 23 | 25
Completed | 22 | 17 | 24
Not Completed | 0 | 6 | 1
Not completed — Non-compliance with facility policies | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Period: Third Intervention
Arm/Group | Guanfacine First | Moxifloxacin First | Placebo First
Started | 22 | 17 | 24
Completed | 21 | 17 | 23
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine First | Moxifloxacin First | Placebo First | Total
Number analyzed (Participants) | 31 | 25 | 27 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 25 | 27 | 83
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (7.55) | 30.8 (10.02) | 30.2 (8.71) | 29.4 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 14 | 43
  Male | 15 | 12 | 13 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 25 | 27 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Electrocardiogram Results (QTcNi) at Time of Maximum Plasma Concentration (Tmax) on Day 1
Description: QTcNi is the QT interval using a subject-specific correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate (e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline, Tmax (time of subject-specific maximum plasma concentration)
Population: Pharmacodynamic (PD) population consists of all evaluable subjects with no major protocol deviations. "Evaluable" subjects were defined as subjects who received a Day 6 dose and had Day 6 data for the primary and secondary endpoints for all three periods.
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Guanfacine 4 mg: 4 mg Immediate-release Guanfacine HCl
- Moxifloxacin: 400 mg Avelox, positive control
Arm/Group | Guanfacine 4 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 57 | 58 | 57 | 58
msec | -3.37 (1.00) [-4.52 to -0.34] | 12.96 (1.03) [11.45 to 16.29] | -0.94 (1.02) | -0.91 (1.04)
Statistical Analysis 1: Comparison: Guanfacine 4 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = -2.43, 90% CI [-4.52 to -0.34]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 13.87, 90% CI [11.45 to 16.29]

2. Primary Outcome: Change From Baseline in Electrocardiogram Results (QTcNi) at Tmax on Day 6
Description: as for outcome 1
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Guanfacine 8 mg: 8 mg Immediate-release Guanfacine HCl
Arm/Group | Guanfacine 8 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 58 | 45 | 58 | 44
msec | -12.45 (1.50) [-11.37 to -4.78] | 8.99 (1.79) [9.33 to 16.93] | -4.37 (1.52) | -4.13 (1.84)
Statistical Analysis 1: Comparison: Guanfacine 8 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = -8.08, 90% CI [-11.37 to -4.78]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 13.13, 90% CI [9.33 to 16.93]

3. Primary Outcome: Change From Baseline in Electrocardiogram Results (QTcF) at Tmax on Day 1
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate (e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Guanfacine 4 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 57 | 58 | 57 | 58
msec | 0.15 (0.96) [-1.07 to 3.03] | 9.96 (0.92) [8.97 to 13.24] | -0.83 (0.97) | -1.14 (0.92)
Statistical Analysis 1: Comparison: Guanfacine 4 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = 0.98, 90% CI [-1.07 to 3.03]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 11.11, 90% CI [8.97 to 13.24]

4. Primary Outcome: Change From Baseline in Electrocardiogram Results (QTcF) at Tmax on Day 6
Description: as for outcome 3
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Guanfacine 8 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 58 | 45 | 58 | 44
msec | -2.67 (1.24) [-0.99 to 4.27] | 6.44 (1.65) [7.63 to 13.97] | -4.31 (1.25) | -4.35 (1.68)
Statistical Analysis 1: Comparison: Guanfacine 8 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = 1.64, 90% CI [-0.99 to 4.27]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 10.80, 90% CI [7.63 to 13.97]

5. Primary Outcome: Change From Baseline in Heart Rate (HR) at Tmax on Day 1
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Guanfacine 4 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 57 | 58 | 57 | 58
bpm | -7.18 (0.58) [-8.01 to -5.51] | 5.46 (0.79) [3.08 to 6.38] | -0.42 (0.58) | 0.73 (0.79)
Statistical Analysis 1: Comparison: Guanfacine 4 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = -6.76, 90% CI [-8.01 to -5.51]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 4.73, 90% CI [3.08 to 6.38]

6. Primary Outcome: Change From Baseline in Heart Rate (HR) at Tmax on Day 6
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Guanfacine 8 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 58 | 45 | 58 | 44
bpm | -19.74 (0.89) [-21.92 to -17.78] | 4.66 (0.83) [1.77 to 5.11] | 0.11 (0.89) | 1.22 (0.85)
Statistical Analysis 1: Comparison: Guanfacine 8 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = -19.85, 90% CI [-21.92 to -17.78]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 3.44, 90% CI [1.77 to 5.11]

7. Primary Outcome: Change From Baseline in Electrocardiogram Results (QT) Interval at Tmax on Day 1
Description: QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate (e.g., the faster the heart rate, the shorter the QT interval).
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Guanfacine 4 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 57 | 58 | 57 | 58
msec | 15.88 (1.63) [11.75 to 18.89] | -1.27 (1.74) [-2.77 to 4.63] | 0.56 (1.63) | -2.20 (1.74)
Statistical Analysis 1: Comparison: Guanfacine 4 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = 15.32, 90% CI [11.75 to 18.89]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 0.93, 90% CI [-2.77 to 4.63]

8. Primary Outcome: Change From Baseline in Electrocardiogram Results (QT) Interval at Tmax on Day 6
Description: as for outcome 7
Time Frame: Baseline and Tmax (time of subject-specific maximum plasma concentration)
Population: PD population
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Guanfacine 8 mg | Moxifloxacin | Placebo (Guanfacine) | Placebo (Moxifloxacin)
Number analyzed (Participants) | 58 | 45 | 58 | 44
msec | 46.21 (2.40) [44.71 to 54.98] | -3.09 (2.15) [-0.41 to 7.66] | -3.63 (2.40) | -6.71 (2.19)
Statistical Analysis 1: Comparison: Guanfacine 8 mg vs Placebo (Guanfacine); Test type: Superiority or Other; Mean Difference (Final Values) = 49.85, 90% CI [44.71 to 54.98]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo (Moxifloxacin); Test type: Superiority or Other; Mean Difference (Final Values) = 3.63, 90% CI [-0.41 to 7.66]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Guanfacine and Moxifloxacin on Day 1
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: Pharmacokinetic (PK) population consists of all subjects in the safety population (subjects who had taken one dose of study medication and had one follow-up safety assessment completed) who had evaluable concentration-time profiles.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Guanfacine 4 mg | Moxifloxacin
Number analyzed (Participants) | 76 | 72
ng/ml | 8.51 (1.77) | 1943.1 (463.8)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Guanfacine and Moxifloxacin on Day 6
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Guanfacine 8 mg | Moxifloxacin
Number analyzed (Participants) | 64 | 57
ng/ml | 24.70 (6.10) | 2003.4 (477.4)

11. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Guanfacine and Moxifloxacin on Day 1
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Guanfacine 4 mg | Moxifloxacin
Number analyzed (Participants) | 76 | 72
hours | 3.9 (1.9) | 2.13 (1.08)

12. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Guanfacine and Moxifloxacin on Day 6
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Guanfacine 8 mg | Moxifloxacin
Number analyzed (Participants) | 64 | 57
hours | 5.2 (2.3) | 1.78 (0.89)

13. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) for Guanfacine and Moxifloxacin on Day 1
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Guanfacine 4 mg | Moxifloxacin
Number analyzed (Participants) | 76 | 72
ng.h/ml | 110.8 (24.4) | 19892 (4670)

14. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) for Guanfacine and Moxifloxacin on Day 6
Time Frame: pre-dose and 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Guanfacine 8 mg | Moxifloxacin
Number analyzed (Participants) | 64 | 57
ng.h/ml | 370.3 (101.3) | 20767 (4396)

ADVERSE EVENTS:
Groups:
- Guanfacine: Immediate-release Guanfacine HCl
- Moxifloxacin: Avelox, positive control
Arm/Group | Guanfacine | Moxifloxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 5/76 | 0/72 | 0/68
Other Adverse Events (participants affected / at risk) | 76/76 | 46/72 | 39/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine (N=76) | Moxifloxacin (N=72) | Placebo (N=68)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine (N=76) | Moxifloxacin (N=72) | Placebo (N=68)
Dry mouth (Gastrointestinal disorders) | 50 | 2 | 0
Dizziness (Nervous system disorders) | 47 | 6 | 5
Asthenia (General disorders) | 43 | 6 | 1
Constipation (Gastrointestinal disorders) | 32 | 4 | 3
Headache (Nervous system disorders) | 23 | 8 | 15
Nausea (Gastrointestinal disorders) | 13 | 14 | 5
Tinnitus (Ear and labyrinth disorders) | 12 | 1 | 0
Vision blurred (Eye disorders) | 10 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 1
Dry eye (Eye disorders) | 8 | 4 | 1
Mucosal dryness (General disorders) | 8 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 7 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 3
Vomiting (Gastrointestinal disorders) | 6 | 4 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 8 | 9
Diarrhea (Gastrointestinal disorders) | 5 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 3
Fatigue (General disorders) | 5 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 5 | 1 | 0
Paresthesia (Nervous system disorders) | 5 | 1 | 0
Scotoma (Eye disorders) | 5 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 0 | 0
Hot flush (Vascular disorders) | 4 | 1 | 1
Hypotension (Vascular disorders) | 4 | 0 | 0
Irritability (General disorders) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually